CLINICAL TRIAL: NCT03992352
Title: Composite Health Assessment Risk Model (CHARM) for Older Adults: Applying Pre-Transplant Comorbidity, Geriatric Assessment, and BioMarkers on Non-Relapse Mortality After Allogeneic Transplant (BMT CTN 1704)
Brief Title: Composite Health Assessment Risk Model (CHARM) for Older Adults (BMT CTN 1704)
Acronym: BMT CTN 1704
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: BMT CTN 1704; 5U24HL138660-02 (NIH)
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Age 60+ with planned HCT for Hematologic Malignancy: Subjects 60 years or older with a planned allogeneic transplantation for a hematologic malignancy.
  Interventions: Diagnostic Test: Age 60+ with planned HCT for Hematologic Malignancy

INTERVENTIONS:
Diagnostic Test: Age 60+ with planned HCT for Hematologic Malignancy — questionnaires, geriatric assessments

SUMMARY:
Prospective observational multicenter study of allogeneic Hematopoietic Stem Cell Transplantation (HCT) in recipients 60 years and older to assess important determinants of health status to be combined into a composite health risk model to improve risk assessment of non-relapse mortality (NRM).

DETAILED DESCRIPTION:
At baseline, standardized Geriatric Assessment (GA) tools incorporating subject reported data and bedside testing will be collected. HCT-Comorbidity Index (CI) scores will be assigned and C-reactive protein (CRP) and albumin will be measured locally. Serial measures at 3, 6, and 12 months for frailty, skilled facility admission, and quality of life (QOL) using PROMIS measures for physical function, depression and anxiety will be determined. Graft Versus Host Disease (GVHD) through one year, serious toxicities through day 100, cognitive status at day 100 and causes of death will be captured.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 60.0 years old at time of enrollment.
2. Hematological malignancy as an indication for allogeneic transplantation.
3. Eligible for allogeneic transplantation based on institutional standards
4. First allogeneic transplant planned. Any conditioning regimen and allogeneic donor is acceptable.
5. Able to speak and read English. Spanish, and Mandarin will be acceptable when sites have ability to perform healthcare provider tests in those languages.
6. Written informed consent

Exclusion Criteria:

1. Prior allogeneic HCT

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 60+ receiving first allogeneic Hematopoetic Cell Transplantation for a hematologic malignancy
Sampling Method: Probability Sample
Enrollment: 1229 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
One Year Non-Relapse Mortality | 1 year
  To determine the set of assessments and biomarkers that could together constitute a robust and valid composite health risk model for accurate personalized estimation of NRM by analyzing data collected from all measures pre and post transplant.

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival
Cumulative Incidence of Frailty | 1 Year
  Cumulative Incidence of Frailty determined by score determined through the Hopkins Frailty Phenotype assessment on a scale of 0-5 where a score of 3 or more is considered 'frail'.
Cumulative incidence of disability | 1 Year
  Cumulative incidence of disability measured through Lawton instrumental activities of daily living (IADL) assessment. Disability is defined as any assistance needed for a specific IADL domain, and measured by a worsening of disability score by one or more IADL within one year.
Cumulative incidence of admission to a skilled nursing facility | 1 Year
  Cumulative incidence of admission to a skilled nursing facility
HRQOL using PROMIS domains | 1 Year
  Health Related Quality of Life as measured using the PROMIS Global Health Physical Function, Anxiety, and Depression domains on scales from 0-100 where 50 is the mean score in a healthy reference population. A higher score indicates 'more' of that domain - for this study that would be more physical function, more anxiety, or more depression than the reference population.
Cumulative incidence of serious organ toxicity by day 100 | 100 Days
  Cumulative incidence of serious organ toxicity by day 100
Cumulative incidence of acute grade 2-4 GVHD | 100 days
  Cumulative incidence of acute grade 2-4 GVHD at 100 days, 6 months and 1 year and chronic GVHD requiring treatment with systemic immune-suppression at 6 months and 1 year
Cumulative incidence of acute grade 2-4 GVHD | 6 months
  Cumulative incidence of acute grade 2-4 GVHD at 100 days, 6 months and 1 year and chronic GVHD requiring treatment with systemic immune-suppression at 6 months and 1 year
Cumulative incidence of acute grade 2-4 GVHD | 1 year
  Cumulative incidence of acute grade 2-4 GVHD at 100 days, 6 months and 1 year and chronic GVHD requiring treatment with systemic immune-suppression at 6 months and 1 year
Chronic GVHD requiring treatment with systemic immune-suppression | 6 months
  Cumulative incidence of acute grade 2-4 GVHD at 100 days, 6 months and 1 year and chronic GVHD requiring treatment with systemic immune-suppression at 6 months and 1 year
Chronic GVHD requiring treatment with systemic immune-suppression | 1 year
  Cumulative incidence of acute grade 2-4 GVHD at 100 days, 6 months and 1 year and chronic GVHD requiring treatment with systemic immune-suppression at 6 months and 1 year
Survival after development of acute grade 2-4 GVHD | 1 year
  Survival after development of acute grade 2-4 GVHD
Cognitive decline at day 100 | Day 100
  Cognitive decline at day 100 as measured using the Montreal Cognitive Assessment (MoCA) as a rapid screening instrument for mild genitive dysfunction. MoCA uses a scale of 0-30 where 26-30 indicates the normal range in healthy populations. Cognitive decline will be defined as a 2 point or greater decline from baseline on total score.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, MS, Principal Investigator — City of Hope Medical Center; Mohamed Sorror, MD, MSc, Principal Investigator — Fred Hutchinson Cancer Center; Wael Saber, MD, MS, Study Chair — Medical College of Wisconsin/CIBMTR
Locations (50):
- United States (50):
  - Mayo Clinic Arizona and Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - University of Florida, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana Blood and Marrow Transplantation, Beech Grove, Indiana
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Blood and Marrow Transplant Program, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Hospital Bone Marrow Transplant Program, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Medicine, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Siedman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State Universtiy, Columbus, Ohio
  - HCA Health Services of Oklahoma, Inc., University of OK, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospitals, Inc., Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pidala J, Craig BM, Lee SJ, Majhail N, Quinn G, Anasetti C. Practice variation in physician referral for allogeneic hematopoietic cell transplantation. Bone Marrow Transplant. 2013 Jan;48(1):63-7. doi: 10.1038/bmt.2012.95. Epub 2012 Jun 18. PMID 22705801
- [Background] Appelbaum FR, Anasetti C, Antin JH, Atkins H, Davies S, Devine S, Giralt S, Heslop H, Laport G, Lee SJ, Logan B, Pasquini M, Pulsipher M, Stadtmauer E, Wingard JR, Horowitz MM. Blood and marrow transplant clinical trials network state of the Science Symposium 2014. Biol Blood Marrow Transplant. 2015 Feb;21(2):202-24. doi: 10.1016/j.bbmt.2014.10.003. Epub 2014 Oct 15. No abstract available. PMID 25445636
- [Background] Juliusson G, Lazarevic V, Horstedt AS, Hagberg O, Hoglund M; Swedish Acute Leukemia Registry Group. Acute myeloid leukemia in the real world: why population-based registries are needed. Blood. 2012 Apr 26;119(17):3890-9. doi: 10.1182/blood-2011-12-379008. Epub 2012 Mar 1. PMID 22383796
- [Background] Mrozek K, Marcucci G, Nicolet D, Maharry KS, Becker H, Whitman SP, Metzeler KH, Schwind S, Wu YZ, Kohlschmidt J, Pettenati MJ, Heerema NA, Block AW, Patil SR, Baer MR, Kolitz JE, Moore JO, Carroll AJ, Stone RM, Larson RA, Bloomfield CD. Prognostic significance of the European LeukemiaNet standardized system for reporting cytogenetic and molecular alterations in adults with acute myeloid leukemia. J Clin Oncol. 2012 Dec 20;30(36):4515-23. doi: 10.1200/JCO.2012.43.4738. Epub 2012 Sep 17. PMID 22987078
- [Background] Burnett AK, Russell NH, Hills RK, Kell J, Nielsen OJ, Dennis M, Cahalin P, Pocock C, Ali S, Burns S, Freeman S, Milligan D, Clark RE. A comparison of clofarabine with ara-C, each in combination with daunorubicin as induction treatment in older patients with acute myeloid leukaemia. Leukemia. 2017 Feb;31(2):310-317. doi: 10.1038/leu.2016.225. Epub 2016 Sep 2. PMID 27624670
- [Background] Rashidi A, Ebadi M, Colditz GA, DiPersio JF. Outcomes of Allogeneic Stem Cell Transplantation in Elderly Patients with Acute Myeloid Leukemia: A Systematic Review and Meta-analysis. Biol Blood Marrow Transplant. 2016 Apr;22(4):651-657. doi: 10.1016/j.bbmt.2015.10.019. Epub 2015 Oct 31. PMID 26529178
- [Background] Devine SM, Owzar K, Blum W, Mulkey F, Stone RM, Hsu JW, Champlin RE, Chen YB, Vij R, Slack J, Soiffer RJ, Larson RA, Shea TC, Hars V, Sibley AB, Giralt S, Carter S, Horowitz MM, Linker C, Alyea EP. Phase II Study of Allogeneic Transplantation for Older Patients With Acute Myeloid Leukemia in First Complete Remission Using a Reduced-Intensity Conditioning Regimen: Results From Cancer and Leukemia Group B 100103 (Alliance for Clinical Trials in Oncology)/Blood and Marrow Transplant Clinical Trial Network 0502. J Clin Oncol. 2015 Dec 10;33(35):4167-75. doi: 10.1200/JCO.2015.62.7273. Epub 2015 Nov 2. PMID 26527780
- [Background] Muffly L, Pasquini MC, Martens M, et al. Increasing Use of Allogeneic Hematopoietic Cell Transplantation (HCT) in Patients Age 70 Years and Older: A CIBMTR Study of Trends and Outcomes. Biology of Blood and Marrow Transplant.22:S68-S69.
- [Background] Blaise D, Furst S, Crocchiolo R, El-Cheikh J, Granata A, Harbi S, Bouabdallah R, Devillier R, Bramanti S, Lemarie C, Picard C, Chabannon C, Weiller PJ, Faucher C, Mohty B, Vey N, Castagna L. Haploidentical T Cell-Replete Transplantation with Post-Transplantation Cyclophosphamide for Patients in or above the Sixth Decade of Age Compared with Allogeneic Hematopoietic Stem Cell Transplantation from an Human Leukocyte Antigen-Matched Related or Unrelated Donor. Biol Blood Marrow Transplant. 2016 Jan;22(1):119-24. doi: 10.1016/j.bbmt.2015.08.029. Epub 2015 Sep 1. PMID 26341397
- [Background] Kasamon YL, Bolanos-Meade J, Prince GT, Tsai HL, McCurdy SR, Kanakry JA, Rosner GL, Brodsky RA, Perica K, Smith BD, Gladstone DE, Swinnen LJ, Showel MM, Matsui WH, Huff CA, Borrello I, Pratz KW, McDevitt MA, Gojo I, Dezern AE, Shanbhag S, Levis MJ, Luznik L, Ambinder RF, Fuchs EJ, Jones RJ. Outcomes of Nonmyeloablative HLA-Haploidentical Blood or Marrow Transplantation With High-Dose Post-Transplantation Cyclophosphamide in Older Adults. J Clin Oncol. 2015 Oct 1;33(28):3152-61. doi: 10.1200/JCO.2014.60.4777. Epub 2015 Aug 10. PMID 26261255
- [Background] Sandhu KS, Brunstein C, DeFor T, Bejanyan N, Arora M, Warlick E, Weisdorf D, Ustun C. Umbilical Cord Blood Transplantation Outcomes in Acute Myelogenous Leukemia/Myelodysplastic Syndrome Patients Aged >/=70 Years. Biol Blood Marrow Transplant. 2016 Feb;22(2):390-393. doi: 10.1016/j.bbmt.2015.09.020. Epub 2015 Sep 28. PMID 26415559
- [Background] Basak GW, Sánchez-Ortega I, Beohou E, et al. Allogeneic Hematopoietic Cell Transplantation in Elderly Patients Aged 65 and Older: A Retrospective Analysis By the Complications and Quality of Life Working Party of the EBMT. Blood. 2016;128:681-681.
- [Background] Soto-Perez-de-Celis E, Li D, Yuan Y, Lau YM, Hurria A. Functional versus chronological age: geriatric assessments to guide decision making in older patients with cancer. Lancet Oncol. 2018 Jun;19(6):e305-e316. doi: 10.1016/S1470-2045(18)30348-6. Epub 2018 Jun 1. PMID 29893262
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- [Background] Sorror ML, Logan BR, Zhu X, Rizzo JD, Cooke KR, McCarthy PL, Ho VT, Horowitz MM, Pasquini MC. Prospective Validation of the Predictive Power of the Hematopoietic Cell Transplantation Comorbidity Index: A Center for International Blood and Marrow Transplant Research Study. Biol Blood Marrow Transplant. 2015 Aug;21(8):1479-87. doi: 10.1016/j.bbmt.2015.04.004. Epub 2015 Apr 7. PMID 25862591
- [Background] Raimondi R, Tosetto A, Oneto R, Cavazzina R, Rodeghiero F, Bacigalupo A, Fanin R, Rambaldi A, Bosi A. Validation of the Hematopoietic Cell Transplantation-Specific Comorbidity Index: a prospective, multicenter GITMO study. Blood. 2012 Aug 9;120(6):1327-33. doi: 10.1182/blood-2012-03-414573. Epub 2012 Jun 27. PMID 22740454
- [Background] Sorror ML, Storb RF, Sandmaier BM, Maziarz RT, Pulsipher MA, Maris MB, Bhatia S, Ostronoff F, Deeg HJ, Syrjala KL, Estey E, Maloney DG, Appelbaum FR, Martin PJ, Storer BE. Comorbidity-age index: a clinical measure of biologic age before allogeneic hematopoietic cell transplantation. J Clin Oncol. 2014 Oct 10;32(29):3249-56. doi: 10.1200/JCO.2013.53.8157. Epub 2014 Aug 25. PMID 25154831
- [Background] Muffly LS, Kocherginsky M, Stock W, Chu Q, Bishop MR, Godley LA, Kline J, Liu H, Odenike OM, Larson RA, van Besien K, Artz AS. Geriatric assessment to predict survival in older allogeneic hematopoietic cell transplantation recipients. Haematologica. 2014 Aug;99(8):1373-9. doi: 10.3324/haematol.2014.103655. Epub 2014 May 9. PMID 24816237
- [Background] Alousi AM, Le-Rademacher J, Saliba RM, Appelbaum FR, Artz A, Benjamin J, Devine SM, Kan F, Laughlin MJ, Lazarus HM, Liesveld J, Perales MA, Maziarz RT, Sabloff M, Waller EK, Eapen M, Champlin RE. Who is the better donor for older hematopoietic transplant recipients: an older-aged sibling or a young, matched unrelated volunteer? Blood. 2013 Mar 28;121(13):2567-73. doi: 10.1182/blood-2012-08-453860. Epub 2013 Jan 29. PMID 23361908
- [Background] Muffly LS, Boulukos M, Swanson K, Kocherginsky M, Cerro PD, Schroeder L, Pape L, Extermann M, Van Besien K, Artz AS. Pilot study of comprehensive geriatric assessment (CGA) in allogeneic transplant: CGA captures a high prevalence of vulnerabilities in older transplant recipients. Biol Blood Marrow Transplant. 2013 Mar;19(3):429-34. doi: 10.1016/j.bbmt.2012.11.006. Epub 2012 Nov 15. PMID 23160006
- [Background] Masnoon N, Shakib S, Kalisch-Ellett L, Caughey GE. What is polypharmacy? A systematic review of definitions. BMC Geriatr. 2017 Oct 10;17(1):230. doi: 10.1186/s12877-017-0621-2. PMID 29017448
- [Background] Hurria A, Cirrincione CT, Muss HB, Kornblith AB, Barry W, Artz AS, Schmieder L, Ansari R, Tew WP, Weckstein D, Kirshner J, Togawa K, Hansen K, Katheria V, Stone R, Galinsky I, Postiglione J, Cohen HJ. Implementing a geriatric assessment in cooperative group clinical cancer trials: CALGB 360401. J Clin Oncol. 2011 Apr 1;29(10):1290-6. doi: 10.1200/JCO.2010.30.6985. Epub 2011 Feb 28. PMID 21357782
- [Background] Hurria A, Mohile S, Gajra A, Klepin H, Muss H, Chapman A, Feng T, Smith D, Sun CL, De Glas N, Cohen HJ, Katheria V, Doan C, Zavala L, Levi A, Akiba C, Tew WP. Validation of a Prediction Tool for Chemotherapy Toxicity in Older Adults With Cancer. J Clin Oncol. 2016 Jul 10;34(20):2366-71. doi: 10.1200/JCO.2015.65.4327. Epub 2016 May 16. PMID 27185838
- [Background] Holmes HM, Des Bordes JK, Kebriaei P, Yennu S, Champlin RE, Giralt S, Mohile SG. Optimal screening for geriatric assessment in older allogeneic hematopoietic cell transplantation candidates. J Geriatr Oncol. 2014 Oct 1;5(4):422-30. doi: 10.1016/j.jgo.2014.04.004. Epub 2014 May 14. PMID 24835889
- [Background] Olin RL, Andreadis C, Martin TG, et al. Comprehensive Geriatric Assessment Identifies Significant Functional Impairments in Older Hematopoietic Cell Transplant Recipients. Biology of Blood and Marrow Transplant.20:S65-S66.
- [Background] Wood WA, Deal AM, Reeve BB, Abernethy AP, Basch E, Mitchell SA, Shatten C, Hie Kim Y, Whitley J, Serody JS, Shea T, Battaglini C. Cardiopulmonary fitness in patients undergoing hematopoietic SCT: a pilot study. Bone Marrow Transplant. 2013 Oct;48(10):1342-9. doi: 10.1038/bmt.2013.58. Epub 2013 Apr 15. PMID 23584437
- [Background] Jones LW, Devlin SM, Maloy MA, Wood WA, Tuohy S, Espiritu N, Aquino J, Kendig T, Michalski MG, Gyurkocza B, Schaffer WL, Ali B, Giralt S, Jakubowski AA. Prognostic Importance of Pretransplant Functional Capacity After Allogeneic Hematopoietic Cell Transplantation. Oncologist. 2015 Nov;20(11):1290-7. doi: 10.1634/theoncologist.2015-0200. Epub 2015 Oct 7. PMID 26446235
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Derived] Artz AS, Logan BR, Saber W, Geller N, Bellach A, Kou J, Wood WA, McCarty J, Knight TG, Runaas L, Johnston L, Walston JD, Nakamura R, Mishra A, Uberti J, Dahi PB, Saultz JN, McCurdy SR, Morris LE Jr, Imus P, Hogan WJ, Nadiminti KV, Bhatt VR, Olin RL, Maakaron JE, Sobecks RM, Wall SA, Mattila D, Protz B, Devine SM, Horowitz MM, Sorror ML. CHARM is Prognostic of Geriatric Morbidity and Toxicity after Allogeneic Transplant for Older Adults: BMT CTN 1704 Study. Blood Adv. 2025 Nov 21:bloodadvances.2025018340. doi: 10.1182/bloodadvances.2025018340. Online ahead of print. PMID 41269781
- [Derived] Sorror ML, Saber W, Logan B, Geller N, Bellach A, Kou J, Wood W, McCarty JM, Knight TG, Runaas L, Johnston L, Walston J, Nakamura R, Jarrett L, Mishra A, Uberti J, Dahi PB, Saultz JN, McCurdy SR, Morris LE, Imus PH, Hogan WJ, Nadiminti K, Bhatt VR, Olin R, Maakaron J, Sobecks R, Wall SA, Mattila D, Protz B, Devine SM, Horowitz MM, Artz AS. Novel composite health assessment risk model for older allogeneic transplant recipients: BMT-CTN 1704. Blood Adv. 2025 Jul 8;9(13):3268-3280. doi: 10.1182/bloodadvances.2025015793. PMID 40101246

DOCUMENTS (1):
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT03992352/ICF_000.pdf